CLINICAL TRIAL: NCT04746716
Title: Long Term Results of Psychoeducation and Cognitive Rehabilitation After Mild Traumatic Brain Injury
Acronym: ReLoT-TCCL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201206
Record Dates: First submitted 2020-11-19; First posted 2021-02-10 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Mild Traumatic Brain Injury
Keywords: mTBI; prognosis; rehabilitation; long term results
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Psychoeducation and Cognitive Rehabilitation After Mild Traumatic Brain Injury: Patient who had a psychoeducation and Cognitive Rehabilitation After their Mild Traumatic Brain Injury
  Interventions: Other: Phone call
- No Psychoeducation and Cognitive Rehabilitation After Mild Traumatic Brain Injury: Patient who hadn't a psychoeducation and Cognitive Rehabilitation After their Mild Traumatic Brain Injury
  Interventions: Other: Phone call

INTERVENTIONS:
Other: Phone call — Phone call to the patient to complete quality of life scales

SUMMARY:
Mild traumatic brain injury (mTBI) accounts for 70-90% of brain injuries, with 600 cases of mTBI per 100 000 people in the united states, but only 100-300 mTBI patients per 100 000 people receive hospital-based care. Symptoms reported immediately after injury tend to diminish over the following 10 days and are generally resolved by 3 months. However, in 15-25% of cases , problems persist, and may even worsen, at 3 months. Physical, emotional, and behavioral factors can be affected. Physical disorders include pain and fatigue. Sleep disorders are also common. Persistent symptoms can affect patient outcomes (affecting all aspects of life) and increase public healthcare costs .In a previous study (NCT03811626, Efficacy of Psychoeducation and Cognitive Rehabilitation After Mild Traumatic Brain Injury for Preventing Post-concussional Syndrome in Individuals With High Risk of Poor Prognosis: A Randomized Clinical Trial. The investigators were able to demonstrate that early multidisciplinary management improved the outcome and prognosis of patients by statistically significantly reducing the percentage of patients with Post traumatic syndrome distress at six months (6% for the treated group versus 52% for the control group, p < 0.001).

It seems important to verify that if this short-term improvement (6 months after the trauma) persists in the long term, and therefore at a distance from the end of the initially proposed rehabilitation.

DETAILED DESCRIPTION:
80 mTBI patients included in the previous study (NCT03811626) will be contacted by phone and an assessment consisting of questionnaires (QOLIBRI, SF-36, Posttraumatic stress disorder Checklist Scale (PCLS ) , ProQol) will be offered to them.

ELIGIBILITY:
Inclusion Criteria:

* all patients from our previous study NCT03811626 and included by our center
* Patient informed and willing to participate

Exclusion Criteria:

* Patient without social security

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 mild traumatic brain injured patients included in our previous study (NCT03811626)will be contacted by phone
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-03-02 (Estimated); Primary Completion 2021-09-02 (Estimated); Study Completion 2021-09-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the long term results of Psychoeducation and Cognitive Rehabilitation After Mild Traumatic Brain Injury | At inclusion = Day 1
  quality of life questionnaire QOLIBRI (Quality of Life after Brain Injury). The QOLIBRI is a comprehensive questionnaire with 37 items covering six dimensions to assess health-related quality of life. Each items has to ba scaled from 1 (Not at all affected) to 5 (Very).The subscale scores can be used separately, or can be combined to give a profile of quality of life. All item responses can also be summed to give a total score.

SECONDARY OUTCOMES:
Contribution of knowledge on the epidemiology of Mild Traumatic Brain Injury | At inclusion = Day 1
  quality of life questionnaire SF-36 : The 36-Item Short Form Survey (SF-36) is an oft-used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study[1].
  It comprises 36 questions which cover eight domains of health. Scores for the different domains are converted and pooled using a scoring key, for a total score indicating a range of low to high quality of life
Contribution of knowledge on the epidemiology of Mild Traumatic Brain Injury | At inclusion = Day 1
  PCLS (Posttraumatic Stress Disorder Checklist Scale). 17 items rated from 1 (never) to 5 (Very often)
Contribution of knowledge on the epidemiology of Mild Traumatic Brain Injury | At inclusion = Day 1
  Professional Quality of Life Scale : The ProQOL has sub-scales for compassion satisfaction, burnout and compassion fatigue. There are 30questions rated from 1(Never) to 5(Very often)

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No